CLINICAL TRIAL: NCT00381758
Title: A Randomized, Double-Blind Comparison of the Time Course of Response to Two Extended-Release Oral Delivery Systems for Methylphenidate in Pediatric Patients With Attention Deficit Hyperactivity Disorder in an Analog Classroom Setting: The CoMACS Study
Brief Title: The COMACS Study: A Comparison of Methylphenidates in an Analog Classroom Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CD00600
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Methylphenidate; Metadate CD; Concerta; COMACS; Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: Methylphenidate Extended Release Capsules

SUMMARY:
This study was designed to compare Concerta Extended Release tablets with Metadate CD capsules in children with ADHD who were between 6 and 12 years old. The effects on ADHD symptoms, and any side effects of treatment, were measured for 12 hours after dosing in a simulated classroom. The treatments were blinded and the effects were compared with a Placebo.

ELIGIBILITY:
Inclusion Criteria:

* 6 -12 years of age, inclusive
* Have a diagnosis of ADHD
* Receiving an approved form of MPH (methylphenidate) and have demonstrated clinical improvement during this treatment.

Exclusion Criteria:

* IQ below 80.
* The patient, or a first-degree relative, has a confirmed diagnosis of Tourette's syndrome or a clinically significant tic disorder.
* History of seizures (excluding uncomplicated childhood febrile seizures).
* Myocardial infarction within 3 months of study entry, or has a history of cardiac disease, congenital cardiac abnormality, glaucoma, hyperthyroidism.
* Comorbid psychiatric diagnosis.
* Exhibits extreme aggressive behavior or destruction of property, marked anxiety, tension, or agitation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184
Dates: Start 2002-05; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
School Day Efficacy
SKAMP (Swanson Kotkin Agler MFlynn Pelham) ADHD Rating Scale: Deportment Items
1.5 - 7.5 hours post-dosing

SECONDARY OUTCOMES:
SKAMP Attention Items, 1.5-12 hrs;
PERMP (Permanent Product of arithmetic) (# Problems Attempted & # Complete), 1.5-12 hrs;
SNAP IV (Swanson Nolan Pelham), day 3 & 7;
Treatment Emergent Adverse Events, once weekly;
Barkley Symptom scale, once weekly
Patient Satisfaction,once weekly
Parent Satisfaction & Treatment Preference once weekly

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatch, Study Director — UCB Pharma